CLINICAL TRIAL: NCT02161016
Title: A Radiographic and Clinical Outcomes Study Evaluating map3® Cellular Allogeneic Bone Graft in Patients Undergoing Bone Grafting in the Foot/Ankle
Brief Title: A Clinical Study of Outcomes in Foot and Ankle Bone Grafting Using map3® Cellular Allogeneic Bone Graft
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: RTI Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: map3-2014
Record Dates: First submitted 2014-06-06; First posted 2014-06-11 (Estimated); Results first posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-02

CONDITIONS: Foot Deformities, Acquired; Disorder of Joint of Foot; Fracture of Foot; Deformity of Bone
MeSH Terms: conditions — Foot Deformities, Acquired

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- map3 allogeneic bone graft (Other): Patients will receive map3® Cellular Allogeneic Bone Graft containing donor matched stem cells.
  Interventions: Device: map3

INTERVENTIONS:
Device: map3 — Patients will receive map3® Cellular Allogeneic Bone Graft containing donor matched stem cells.

SUMMARY:
This is a single arm pilot study in patients requiring surgical fusion in the foot or ankle. Patients will receive map3® Cellular Allogeneic Bone Graft containing donor matched stem cells. This cohort study will enroll 24 patients total at 1 site. After subjects have signed an informed consent, the baseline visit and examinations will be completed. Patients will be evaluated at 2 weeks, 6 weeks, 3 months, 6 months, 12 months, and 24 months after surgery.

DETAILED DESCRIPTION:
map3® Cellular Allogeneic Bone Graft provides the desired osteoconductive, osteoinductive and osteogenic potential capacities which are essential to optimal fracture healing when bone grafts are implanted. It offers viable MAPC-class cells on a scaffold comprised of demineralize bone matrix (DBM) and cortical cancellous chips. map3® Cellular Allogeneic Bone Graft is considered an allograft, and as such, is indicated for bone repair for orthopaedic indications where autograft is employed. The primary goal of this study is to evaluate the outcomes in bone grafts of the foot or ankle using a stem cell modified allograft (map3® Cellular Allogeneic Bone Graft). The study endpoints will be objectively determined via x-rays and CT scan to assess bony fusion, extremity evaluation using the AFAS and subjective patient scores for foot disabilities and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects will be limited to patients with foot/ankle pathologies requiring fusion, which include midfoot, hindfoot, ankle, double and triple arthrodesis using open surgical technique with supplemental bone graft substitute.
* Life expectancy of at least twenty four (24) months
* Ability to give written informed consent
* All subjects will have a minimum age of eighteen (18) years and a maximum of eighty (80) years.
* Both male and non-pregnant female subjects will be included.
* To facilitate follow-up, study subjects will be limited to the local geographic area of the study site and must be willing to use the rehabilitation facility and physical therapy schedule assigned by the surgeon.
* All subjects must be able to read, write, and comprehend instructions and guidelines in English and understand (and sign as an acknowledgment of their understanding) an informed consent declaration

Exclusion Criteria:

* Patients who have been diagnosed with Charcot foot
* Patients requiring osteotomies or undergoing a revision surgery for non-union
* Patients with additional lower limb injuries requiring concomitant procedures not related to the current foot/ankle procedure
* Patients with soft tissue compromise involving open and/or infected wounds on the study limb
* Patients requiring any other bone grafting product other than study product (map3® Cellular Allogeneic Bone Graft) e.g. rhBMP2 (recombinant human bone morphogenetic protein 2).
* Patients with confirmed diagnosis of abnormal lower limb vasculature or peripheral vascular disease
* Patients with a high Body Mass Index ( BMI > 35)
* Diagnosis of osteonecrosis, metabolic bone diseases or gout
* Diabetic patients who are insulin dependent
* Patients who have received any treatment within the past 12 months which may interfere with bone metabolism (bisphosphonates and/or calcitonin).
* Patients using glucocorticoids > 10 mg/day
* Chronic use (≥ 90 days) of non-steroidal anti-inflammatory drugs (NSAIDS)
* Patients with active cancer or a history of any cancer
* Known allergies to Dimethyl Sulfoxide (DMSO) and/or Human Serum Albumin (HSA)
* Pregnant or lactating females or who are capable of reproduction and will not take acceptable measures to prevent reproduction during the study
* Patients who have tested positive for HTLV, HIV, hepatitis B or hepatitis C, have rheumatoid arthritis, an autoimmune disease or are on chronic immunosuppressive medications
* Require chronic use (≥ 90 days) of anticoagulation therapy
* Active smokers unwilling to comply with surgeons instructions to stop smoking seven (7) days prior to surgery through three (3) month post-op visit
* History of alcohol or drug abuse within 90 days of screening
* Patients currently enrolled or have been enrolled in clinical studies evaluating investigational devices, pharmaceuticals or biologics within 90 days of enrollment.
* Patients unable to give written informed consent and any vulnerable patient population
* Inability to comply with all requirements of this investigation, as well as follow the instructions of the physician

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Radnay, MD, Principal Investigator — Saint Francis Hospital
Locations (1):
- Saint Francis Hospital, Roslyn, New York, United States

REFERENCES:
- [Background] Guyton GP, Miller SD. Stem cells in bone grafting: Trinity allograft with stem cells and collagen/beta-tricalcium phosphate with concentrated bone marrow aspirate. Foot Ankle Clin. 2010 Dec;15(4):611-9. doi: 10.1016/j.fcl.2010.09.003. PMID 21056860
- [Background] Clements JR. Use of allograft cellular bone matrix in multistage talectomy with tibiocalcaneal arthrodesis: a case report. J Foot Ankle Surg. 2012 Jan-Feb;51(1):83-6. doi: 10.1053/j.jfas.2011.09.002. Epub 2011 Oct 20. PMID 22014833

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | map3 Allogeneic Bone Graft
Started | 1
Completed | 0
Not Completed | 1
Not completed — withdrawn by IRB | 1

BASELINE CHARACTERISTICS:
Arm/Group | map3 Allogeneic Bone Graft
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: AOFAS Foot-and-Ankle Score
Description: The American Orthopaedic Foot and Ankle Society score returns an indexed score, from 0 - 100, to assess clinical outcomes following foot /ankle surgery.
Time Frame: 24 months
Arm/Group | map3 Allogeneic Bone Graft
Number analyzed (Participants) | 0

2. Secondary Outcome: SF-36 Score
Description: The SF-36 is a survey for health and well-being.
Time Frame: 24 months
Arm/Group | map3 Allogeneic Bone Graft
Number analyzed (Participants) | 0

3. Secondary Outcome: Foot Ankle Disability Index
Description: The Foot Ankle Disability Index (FADI) is a self-report of function that assesses activities of daily living, with scores ranging from 0 to 100.
Time Frame: 24 months
Arm/Group | map3 Allogeneic Bone Graft
Number analyzed (Participants) | 0

4. Secondary Outcome: CT Scan
Description: A CT scan will be done at 6 months in order to assess bone fusion.
Time Frame: 6 months
Arm/Group | map3 Allogeneic Bone Graft
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Time to Full Weight-bearing
Description: This will be the time from the date of surgery until the patient has full, unassisted weight bearing, and will be measured in weeks.
Time Frame: up to 24 months
Arm/Group | map3 Allogeneic Bone Graft
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | map3 Allogeneic Bone Graft
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less